CLINICAL TRIAL: NCT02882347
Title: The Effect of Somatostatin for Treatment of Post Hepatectomy Liver Failure (PHLF)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Korea University Anam Hospital (Other)
Collaborators: Pharmbio Korea Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Jae Hyun Han, clinical assistant professor, Korea University Anam Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ED15139
Record Dates: First submitted 2016-08-17; First posted 2016-08-29 (Estimated); Last update posted 2016-09-12 (Estimated); Status verified 2016-09

CONDITIONS: Liver Failure
MeSH Terms: conditions — Liver Failure | interventions — Somatostatin

ARMS (1):
- somatostatin group (Experimental): The investigators administrate somatostatin at a rate of 3.5ug/kg/hour to PHLF patients (prothrombin time < 50% and serum total bilirubin > 2.9mg/dl after liver resection) until recovery from liver failure.
  Interventions: Drug: Somatostatin

INTERVENTIONS:
Drug: Somatostatin

SUMMARY:
Post hepatectomy liver failure (PHLF) is a serious medical problem could lead to patient death, however, definite treatment strategy has not been established. The liver is a regenerating organ and the possibility of PHLF could be reduced when the appropriate liver regeneration is guaranteed.

Portal flow has known to be important during liver regeneration. Low portal flow cannot induce proper regeneration, contrary, excessive flow increase shear stress in the hepatic sinusoid resulting liver failure.

Various medications has been used in malignant liver cirrhosis to reduce portal pressure. Among them, somatostatin has been used modulating portal flow reducing portal and sinusoidal pressure.

In this study, the investigators administrate somatostatin at a rate of 3.5ug/kg/hour to PHLF patients (prothrombin time < 50% and serum total bilirubin > 2.9mg/dl after liver resection) until recovery from liver failure. For assessment of the recovery of liver failure, the investigators evaluate aspartate transaminase (AST), alanine transaminase (ALT), serum total bilirubin and prothrombin time periodically after administration of medication.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with PHLF without regard primary disease.
2. Ability to provide written informed consent

Exclusion Criteria:

1. Concomitant surgery for another intraabdominal organs.
2. Severe renal disease requiring dialysis.
3. Patients with coagulation disorders or taking warfarin.
4. Immunosuppressed patients or the patients with autoimmune disorders.
5. Women with pregnant, breast-feeding.
6. Hypersensitivity to somatostatin.
7. Patients treated with other investigational product within 30 days at the consents are obtained.
8. Patients with a significantly reduced cognitive abilities.
9. Not eligible to participate for study at the discretion of investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-07; Primary Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
in hospital mortality | up to 4 weeks

SECONDARY OUTCOMES:
Complication rate | up to 4 weeks
Time to recovery from PHLF (days) | up to 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Sik Kim, Professor, Study Chair — Department of surgery, Korea university Anam hospital
Locations (1):
- Korea university Anam hospital, Seoul, Seoul, South Korea